CLINICAL TRIAL: NCT04415086
Title: Treatment of Patients With COVID-19 With Convalescent Plasma Transfusion: a Multicenter, Open-labeled, Randomized and Controlled Study
Brief Title: Treatment of Patients With COVID-19 With Convalescent Plasma
Acronym: COOPCOVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Ministério da Ciência, Tecnologia, Inovações e Comunicações (Unknown); Faculty of Medicine of Ribeirão Preto (FMRP-USP) (Other); Hospital de Clínicas, Faculdade de Medicina Universidade Estadual de Campinas (Unknown); Hospital Sirio-Libanes (Other); Hospital Israelita Albert Einstein (Other); Grupo Hospitalar Conceição (Other Government); Hospital Ernesto Dornelles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COOP-COVID-19-MCTIC
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; convalescent plasma; efficacy; safety
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 1:1:1 into 3 treatment groups: A- standard (control); B- standard and convalescent plasma in a volume of 200ml (150-300ml); C- standard and convalescent plasma in a volume of 400ml (300-600ml)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Sham Comparator): Participants will receive the standard of care treatment
  Interventions: Biological: convalescent plasma
- Group B (Active Comparator): Participants will receive the standard treatment and convalescent plasma in a volume of 200ml (150-300ml)
  Interventions: Biological: convalescent plasma
- Group C (Active Comparator): Participants will receive the standard treatment and convalescent plasma in a volume of 400ml (300-600ml)
  Interventions: Biological: convalescent plasma

INTERVENTIONS:
Biological: convalescent plasma — The study will be interrupted if the efficacy of the convalescent plasma group is proven, so that all severely ill patients as defined in the study can receive the convalescent plasma treatment. The same will occur if there is no difference in primary outcome with the use of convalescent plasma or serious adverse effects.

SUMMARY:
The COVID-19 pandemic has been spreading continuously, and in Brazil, until May 31, 2020, there have been more than 450.000 cases with more than 28.000 deaths, with daily increases. The present study proposes to evaluate the efficacy and safety of convalescent plasma in treatment of severe cases of COVID-19 in a multicenter, randomized, open-label and controlled study

DETAILED DESCRIPTION:
Eligible patients will be randomized 1:1:1 into 3 treatment groups: A- standard (control); B- standard and convalescent plasma in a volume of 200ml (150-300ml); C- standard and convalescent plasma in a volume of 400ml (300-600ml). The Bayesian multi-arm and multi-stage model will be used, which will allow an interim analysis after the inclusion of 30 patients, with repeated interim analyses for every 30 additional patients. With this, we expect to define not only the efficacy of convalescent plasma, but also the volume of plasma needed if efficacy is proven. The study will be interrupted if the efficacy of the convalescent plasma group is proven, so that all severely ill patients as defined in the study can receive the convalescent plasma treatment. The same will occur if there is no difference in primary outcome with the use of convalescent plasma or serious adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age = or > than 18 years; .
* Laboratory-proven COVID-19 infection by RT-PCR in any clinical sample . Time since symptom onset less than 10 days at the time of screening; - . Presence of COVID-19 pneumonia, with a typical, indeterminate or atypical compatible image in a chest tomography exam (see definition below) -
* Presence of one of the following criteria:
* Need for> 3L of O2 in the catheter / mask or> 25% in the Venturi mask to maintain O2 saturation> 92% B presence of respiratory distress syndrome with PaO2 / FiO2 <300mmHg If intubated, within 48 hours of orotracheal intubation
* Absence of a history of serious adverse reactions to transfusion, for example, anaphylaxis; - .Participation approval by the research clinician

Exclusion Criteria:

* Already enrolled in another clinical trial evaluating antiviral or immunobiological therapy for the treatment of COVID-19.
* IgA deficiency
* Presence of a clinical condition that does not allow infusion of 400 ml of volume at clinical discretion
* Pregnancy or breastfeeding
* Receipt of immunoglobulin in the last 30 days
* Presence of significant risk of death within the next 48 hours at clinical discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Time elapsed until clinical improvement or hospital discharge | Follow up until 28 days after transfusion
  clinical improvement is defined as the time from the randomization date until the decline of 2 categories on the ordinal scale of 10 categories or hospital discharge (whichever comes first)

SECONDARY OUTCOMES:
acute adverse events | Up to 12 hours after transfusion
  incidence of acute adverse events possibly or definitively realted to convalescent plasma transfusion
Clinical Status | "Day 7", "Day 14" and "Day 28"
  Evaluation according to an ordinal scale of 10 categories
Duration of clinical events | Up to 28 days
  Duration of mechanical ventilation, length of hospital stay in survivors up to 28 days and time from the beginning of treatment to death
SARS-CoV-2 in nasopharyngeal swab | Days 0, 1, 3, 7, 14 and 28 after transfusion and control groups
  Detection of SARS-CoV-2 in nasopharyngeal swab
IgG, IgM and IgA titers for SARS-CoV-2 | Days 0, 1, 3, 5, 7, 14 and 28 after transfusion and control groups
  Specific IgG, IgM and IgA titers for SARS-CoV-2
Neutralizing antibodies | 0,1,7 14 and 28 days after transfusion and control groups
  Titers of neutralizing antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Esper G Kallás, PhD, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo - General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song ATW, Rocha V, Mendrone-Junior A, Calado RT, De Santis GC, Benites BD, Costa-Lima C, Vargas T, Marques LS, Fernandes JC, Breda FC, Wendel S, Fachini R, Rizzo LV, Kutner JM, Avelino-Silva VI, Machado RRG, Durigon EL, Chevret S, Kallas EG. Treatment of severe COVID-19 patients with either low- or high-volume of convalescent plasma versus standard of care: A multicenter Bayesian randomized open-label clinical trial (COOP-COVID-19-MCTI). Lancet Reg Health Am. 2022 Jun;10:100216. doi: 10.1016/j.lana.2022.100216. Epub 2022 Mar 15. PMID 35308034

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT04415086/SAP_000.pdf